CLINICAL TRIAL: NCT07289269
Title: Prevalence of Violence Against Infertile Women Attending Infertility Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed hosni dahi hassan, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: violence infertile women
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Infertility Treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Married women with primary or secondary infertility due to male or female factors at reproductive age (18-45 years).

SUMMARY:
Infertility is a major health concern with a great psychosocial impact. It's defined as the inability to achieve pregnancy after 12 months or more of regular unprotected sexual intercourse[1] affecting about 12%-25% of couples in Egypt[2, 3].

People in Egypt prefer extended families to guarantee maintained family line. Therefore, infertility leads to great negative attitudes and extreme pressures on women[4].

Besides the medical advances in the treatment of infertility as a pathological condition, concerted actions should be taken to address the consequences of infertility on other aspects of human wellbeing including violence against infertile women[1].

Infertile women are more vulnerable to depression and stress which are the underlying factors for domestic violence, as they are commonly blamed for this issue. Domestic violence against women is a global public health problem and human rights crime[5]. In 2013, the World Health Organization (WHO) released a report providing global and regional estimates of violence against women, which documented the broad and invasive global prevalence of this problem and its impact on many aspects of women's health[6]. Intimate partner violence is the most common form of violence against women, defined as any form of violence by a current or former male intimate partner that can include emotional/psychological and economic elements in addition to physical and sexual components. In the most recent WHO report on IPV and its consequences for health, The baseline quality of life of the victims of intimate partner violence is significantly impaired when compared with the non-abused controls [7]. the analysis was limited to physical and/or sexual violence because these are the most widely documented manifestations of IPV across studies[8].

This study will be conducted in collaboration with National Women's council and UNFPA Egypt .We are already running a safe women clinic at Women Health Hospital Assiut university since March 2021 aiming to keep women safe and guarding against any type of violence We will conduct this study to evaluate the relation between infertility and violence against Egyptian women. We hypothesized that infertile women would suffer more violance than fertile ones.

ELIGIBILITY:
Inclusion Criteria:

* Married women with primary or secondary infertility due to male or female factors at reproductive age (18-45 years).

Exclusion Criteria:

* • women who refused to participate in the study.

  * Separated or divorced women.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: - Married women with primary or secondary infertility due to male or female factors at reproductive age (18-45 years).
Sampling Method: Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the prevalence violence among women seeking infertility treatment | baseline